CLINICAL TRIAL: NCT03795246
Title: Long-term Follow-up of Sequential Chemotherapy and Stimulation for Fertility Preservation in Young Patients Treated for a Breast Cancer
Brief Title: Follow-up of Sequential Chemotherapy and Stimulation for Fertility Preservation in Young Patients With Breast Cancer
Acronym: KSF2
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Oscar Lambret (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: KSF2-1707
Record Dates: First submitted 2018-12-31; First posted 2019-01-07 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Referral and Consultation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study Process (Experimental): Consultation, Biological Test, Pelvic Ultrasound
  Interventions: Procedure: Consultation; Biological: Biological Test; Procedure: Pelvic Ultrasound

INTERVENTIONS:
Procedure: Consultation — Consultation in oncology: collection of oncological data and ongoing cancer treatments, clinical exam Consultation in gynecology: collection of gynecological data, contraception and reproductive medicine
Biological: Biological Test — Blood test:
  * FSH, LH, E2 and AMH
  * 4 tubes of 7 mL
Procedure: Pelvic Ultrasound — Antral Follicles Count

SUMMARY:
Interventional research with low risks and constraints, prospective and monocentric on the assessment of long-term fertility in patients who underwent an adjuvant sequential chemotherapy with or without a controled ovarian hyperstimulation. This study follows a previous one called NCT 01614704.

DETAILED DESCRIPTION:
The patients will have a follow-up once a year during ten years beginning at the end of their chemotherapy.

They will have a consultation in oncology consisting of:

* a clinical exam,
* a collection and follow-up of oncological data
* a collection of ongoing cancer treatments

and a consultation in gynecology consisting of:

* a pelvic ultrasound scan (for AFC: Antral Follicle Count)
* a biological test (FSH, LH, E2, AMH)
* a collection of gynecological data, contraception and reproductive medicine

ELIGIBILITY:
Inclusion Criteria:

* Patients included in the study CT 01614704
* Informed and written consent
* Affiliated to the National Social Security System

Exclusion Criteria:

* Impossibility to submit at the study procedures due to geographic, social or mental reasons
* Patient deprived of their liberty or under guardianship or tutorship.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 132 (Estimated)
Dates: Start 2018-03-23 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of fertility in terms of cumulative incidence of long-term pregnancy | 10 years after chemotherapy
  for patients who underwent adjuvant sequential chemotherapy of anthracycline and taxane separately, depending on whether or not they have had Controlled Ovarian Hyperstimulation

SECONDARY OUTCOMES:
Assessment of fertility in terms of cumulative incidence of births | 10 years after chemotherapy
  separately, depending on whether or not they have had Controlled Ovarian Hyperstimulation
Assessment of fertility - number of pegnancies spontaneous versus assisted | 10 years after chemotherapy
  describing the pregnancy type - number of pegnancies spontaneous versus assisted, with ot without the use of frozen gametes)
Assessment of fertility - pregnancy outcome : miscarriage or single or multiple birth separately | 10 years after chemotherapy
  describing the pregnancy outcome : miscarriage or single or multiple birth separately, depending on whether or not they have had Controlled Ovarian Hyperstimulation
Assessment of the number of patient willing to re-exploit their frozen gametes | 10 years after chemotherapy
  for patients who have had Controlled Ovarian Hyperstimulation
Assessment of the gonadotoxicity of the adjuvant sequential chemotherapy based on anthracyclines and taxanes - AMH rate | 10 years after chemotherapy
  in terms of AMH rate depending on whether or not they have had Controlled Ovarian Hyperstimulation
Assessment of the gonadotoxicity of the adjuvant sequential chemotherapy based on anthracyclines and taxanes - Antral Follicle Count | 10 years after chemotherapy
  in terms of Antral Follicle Count depending on whether or not they have had Controlled Ovarian Hyperstimulation
Study the long-term carcinologic safety of Controlled Ovarian Hyperstimulation without Letrozole or Tamoxifen co-treatment in terms of survival without relapse | After chemotherapy ad until disease progression or death regardless of the cause, up to 10 years after chemotherapy
  Survival without relapse defined by the time frame between the date of surgery and the date of the first recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Audrey MAILLIEZ, MD, Study Director — Centre Oscar Lambret; Christine DECANTER, MD, Study Director — Centre Hopsitalier Regional Universitaire de Lille - Hôpital Jeanne de Flandre
Locations (1):
- Centre Oscar Lambret, Lille, France